CLINICAL TRIAL: NCT01240954
Title: Comparison of Different Up-dosing Schedules With Osiris
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CA approval not obtained
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OS-I-01
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Allergic Rhinitis
Keywords: Rhinitis; Allergic; Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis | interventions — Osi21 protein, Drosophila

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- OSIRIS (Active Comparator)
  Interventions: Drug: OSIRIS
- OSIRIS other concentration 1 (Experimental)
  Interventions: Drug: OSIRIS other concentration 1
- OSIRIS other concentration 2 (Experimental)
  Interventions: Drug: OSIRIS other concentration 2

INTERVENTIONS:
Drug: OSIRIS — OSIRIS current practice
  Arms: OSIRIS
Drug: OSIRIS other concentration 1 — OSIRIS new concentration 1
  Arms: OSIRIS other concentration 1
Drug: OSIRIS other concentration 2 — OSIRIS new concentration 2
  Arms: OSIRIS other concentration 2

SUMMARY:
The purpose of this study is to compare different up-dosing schedules with Osiris.

ELIGIBILITY:
Inclusion Criteria:

* history of grass pollen allergy
* Positive SPT to grass
* Positive IgE to grass

Exclusion Criteria:

* uncontrolled and severe asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2010-12

PRIMARY OUTCOMES:
evaluate the tolerability of different up-dosing schedules | 30 days

SECONDARY OUTCOMES:
patient's satisfaction | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Krakow, Poland